CLINICAL TRIAL: NCT02089321
Title: Multiplanar Lumbopelvic Control in Patients With Low Back Pain
Status: Completed | Type: Observational
Sponsor: Regis University (Other)
Responsible Party: Principal Investigator, Erika Nelson-Wong, Associate Professor, Regis University
Other Study IDs: NelsonWong_LBP2013
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Low Back Pain
Keywords: low back pain; lumbopelvic assessment; active straight leg raise; active hip abduction
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Low Back Pain: n= 19
  Inclusion Criteria:
  Between the ages of 18 and 70 years Currently seeking, but not yet initiated, treatment from a health care professional (PT, MD, DO, DC) for a chief complaint of pain between the level of the twelfth thoracic vertebrae and the coccyx Able to transition between standing, sitting, supine, prone and sidelying independently
  Exclusion Criteria:
  Signs of neurological impairment including diminished myotatic reflex, sensory impairment or strength deficits in a myotomal pattern No previous spine or hip surgery Serious spinal or systemic pathology Pregnancy within previous 12 months Inability to understand and follow verbal instructions in English
- Healthy Controls: n= 19
  Inclusion Criteria:
  Between the ages of 18 and 70 years No LBP episodes requiring clinical care by a health professional and/or greater than 3 days absence from work/school/recreation within the previous 5 years Able to transition between standing, sitting, supine, prone and sidelying independently
  Exclusion Criteria:
  No previous spine or hip surgery Serious spinal or systemic pathology Pregnancy within previous 12 months Inability to understand and follow verbal instructions in English

SUMMARY:
The purpose of this study was to investigate whether combined assessment of lumbopelvic control during sagittal and frontal plane motion (using two common clinical observational assessments) discriminates between people with and without LBP than single plane assessment alone. It was hypothesized that the two tests used in combination (multiplanar) would perform better than each test used independently (single planar) in accurately discriminating patient cases from healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients with LBP

Inclusion Criteria:

* Age 18-70 years old
* Ability to understand and follow written and verbal instruction in English
* Seeking treatment from a physical therapist for LBP (pain below T12-L1 vertebral segment), prior to initial evaluation (no treatment provided)

Matched Controls: Control subjects will be matched for age, gender, and BMI category to patients with LBP.

Inclusion Criteria:

* Ability to understand and follow written and verbal instruction in English
* No history of LBP during the past 5 years requiring:

  * > 3 day absence from work/school/recreation
  * Clinical Care (MD, DC, DPT, MT) for LBP

Exclusion Criteria:

Patients with LBP

* Pregnancy within past 12 months
* Previous spine or hip surgery
* Serious spinal or systemic pathology
* Inability to transfer from standing to supine to sidelying to prone
* Inability to stand > 20 minutes

Matched Controls

Exclusion Criteria:

* Pregnancy within the past 12 months
* Previous spine or hip surgery
* Inability to transfer from standing to supine to side-lying to prone
* Inability to stand > 20 minutes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with low back pain were recruited from the physical therapy clinic located at Regis University as well as clinical practices from the surrounding area. Control subjects were a community sample.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Performance on Active Hip Abduction Test | Assessed on data collection day
  Examiner scores movement pattern (ability to retain lumbopelvic neutral) during performance of active hip abduction in sidelying using an ordinal scale (0-3) with 0-1 considered a negative test and 2-3 considered a positive test.
Performance on Active Straight Leg Raise Test | Assessed on data collection day
  Participant self-rates degree of difficulty (0-5) to perform active straight leg raise in supine with any non-zero score considered a positive test result.

CONTACTS AND LOCATIONS:
Locations (1):
- Regis University, Denver, Colorado, United States